CLINICAL TRIAL: NCT00962247
Title: Effect of Changing Sedentary Behavior in Youth
Acronym: Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Leonard Epstein, Leonard H. Epstein, Ph.D., State University of New York at Buffalo
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HD039778; 5R01HD039778 (NIH)
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: physical activity; relative reinforcing value; sedentary behavior; obesity
MeSH Terms: conditions — Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sedentary; usual, 25% reduced, 50% reduced (Experimental): The initial 3 weeks of the study, children were asked to maintain their usual targeted sedentary behaviors (TV, video game, computer use) measured by a television reduction device (TV Allowance). The following 3 weeks children were asked to reduce their targeted sedentary behaviors (TV, video game, computer use) by 25% from the usual sedentary condition using a television reduction device (TV Allowance). The final 3 weeks of the study, children were asked to reduce their targeted sedentary behaviors (TV, video game, computer use) by 50% from the usual sedentary condition using a television reduction device (TV Allowance)
  Interventions: Device: Television reduction device

INTERVENTIONS:
Device: Television reduction device — A TV allowance helps turn off the television when the time limits have been met.

SUMMARY:
The primary aim is to examine how reduction in sedentary behaviors influences physical activity and energy intake.

DETAILED DESCRIPTION:
Many youth find television, videos and computer games to be very reinforcing, and they choose to be sedentary rather than physically active. Sedentary behaviors can influence energy balance and body weight by reducing physical activity and increasing energy intake. Research from our laboratory has shown that reducing sedentary behavior can increase physical activity and decrease energy intake, but there is substantial variability in the response of youth to reductions in sedentary behavior. The present proposal is designed to extend our research and explore theoretical models that may help understand why youth vary in their response to increase physical activity when targeted sedentary behaviors are reduced. We hypothesize that the increase in physical activity when sedentary behaviors are reduced is related to the relative reinforcing value (RRV) of physical activity to sedentary behaviors. The RRV of physical activity is a measure of the motivation to be active in youth, and overweight youth who are inactive find physical activity relatively less reinforcing than less overweight youth. We predict that RRV of physical activity will be positively related to the substitution of total physical activity and physical activity in the moderate to vigorous intensity range for sedentary behaviors when targeted sedentary behaviors are reduced. To test this hypothesis, we will study 60 overweight and at risk for overweight 8-12 year-old youth who differ in the RRV of physical activity to sedentary behavior, with equal numbers of boys and girls, in 3 phases: baseline, and reduce television watching from baseline by 25 percent and 50 percent. Each phase will be implemented for three weeks. Order of experimental phases will be counterbalanced across subjects. It is also predicted that reducing sedentary behavior will reduce energy intake and dietary fat intake, and the reduction in energy intake will be greatest for youth with stronger association between eating with television watching and other targeted sedentary behaviors. Liking and outcome expectancy of physical activity will be studied as additional predictors of substitution of physical activity for reductions in sedentary behaviors. Developing a better understanding of why obese youth increase physical activity or decrease energy intake when sedentary behaviors are reduced is important for the treatment of pediatric obesity.

ELIGIBILITY:
Inclusion Criteria:

* above the 85th BMI percentile
* reside in one primary household
* engage in at least 18 hours of sedentary behavior a week

Exclusion Criteria:

* none

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epstein LH, Roemmich JN, Cavanaugh MD, Paluch RA. The motivation to be sedentary predicts weight change when sedentary behaviors are reduced. Int J Behav Nutr Phys Act. 2011 Feb 22;8:13. doi: 10.1186/1479-5868-8-13. PMID 21342518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were recruited from the Buffalo NY area. 460 families were interested in screening for the study with 271 ineligible families, 4 families who were no longer interested and 28 families who withdrew from phone screen, for a total of 157 families eligible for an orientation appointment.
Pre-assignment Details: Prior to enrolling in the protocol, families completed an orientation, at which eligibility and interest were assessed. Families who enrolled, first completed three weeks of monitoring on the Television reduction device to determine eligibility (at least 18 hours/week of screen use) and compliance with physical activity accelerometer use.
Groups:
- Sedentary; Usual, 25% Reduced, 50% Reduced: Children were asked to maintain their usual targeted sedentary behaviors (TV, video game, computer use) measured by a television reduction device (TV Allowance)
Period: Usual Sedentary
Arm/Group | Sedentary; Usual, 25% Reduced, 50% Reduced
Started | 61
Completed | 61
Not Completed | 0
Period: 25% Reduction of Sedentary Activity
Arm/Group | Sedentary; Usual, 25% Reduced, 50% Reduced
Started | 61
Completed | 56
Not Completed | 5
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 1
Period: 50% Reduction of Sedentary Activity
Arm/Group | Sedentary; Usual, 25% Reduced, 50% Reduced
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Sedentary: Children were asked to maintain their usual targeted sedentary behaviors (TV, video game, computer use) measured by a television reduction device (TV Allowance)
Arm/Group | Usual Sedentary
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 42
  More than one race | 8
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: Inches] | 57.4 (3.7)
Weight [Mean (Standard Deviation); unit: lbs] | 118.8 (30.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.0 (4.2)
zBMI [Mean (Standard Deviation); unit: z-score] | 1.8 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: Actigraph activity monitors were used to record physical activity over 3 days, in addition to a weekly physical activity diary. Acti-graph counts were used to estimate energy expenditure during waking hours. Counts per minute describes the average rate of counts, with 0 being at rest and higher numbers indicating more vigorous physical activity.
Time Frame: 3 days
Measure: Mean (Standard Error); unit: counts/minute of physical activity
Groups:
- 25% Sedentary Reduction: Children were asked to reduce their targeted sedentary behaviors (TV, video game, computer use) by 25% from the usual sedentary condition using a television reduction device (TV Allowance)
  Television reduction device: A TV allowance helps turn off the television when the time limits have been met.
- 50% Sedentary Reduction: Children were asked to reduce their targeted sedentary behaviors (TV, video game, computer use) by 50% from the usual sedentary condition using a television reduction device (TV Allowance)
  Television reduction device: A TV allowance helps turn off the television when the time limits have been met.
Arm/Group | Usual Sedentary | 25% Sedentary Reduction | 50% Sedentary Reduction
Number analyzed (Participants) | 56 | 56 | 56
counts/minute of physical activity | 576.9 (23.8) | 572.4 (25.6) | 555.7 (24.3)

2. Secondary Outcome: Energy Intake
Description: Resting metabolic rate was calculated using the activity data from accelerometer (Actigraph) collection. Resting metabolic rate was used to calculate estimated daily energy expenditure. Daily energy expenditure and weight change over the study period was used to estimate energy intake. If weight was stable of the nine weeks, assume energy intake = energy expenditure. A gain of a pound was estimated as equivalent to a positive balance of 3500 calories and a loss of a pound was estimated as equivalent to a negative balance of 3500 calories.
Time Frame: 3 days
Measure: Mean (Standard Error); unit: calories/day
Arm/Group | Usual Sedentary | 25% Sedentary Reduction | 50% Sedentary Reduction
Number analyzed (Participants) | 56 | 56 | 56
calories/day | 2106.4 (65.7) | 2173.5 (65.2) | 2144.3 (74.6)

ADVERSE EVENTS:
Arm/Group | Usual Sedentary
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No